CLINICAL TRIAL: NCT03444532
Title: Feasibility Study of a Randomized Controlled Trial Testing a Sleep Intervention in Prostate Cancer Patients With Insomnia
Brief Title: Feasibility Study Testing a Sleep Intervention in Prostate Cancer Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Christoffer Johansen, Professor, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sleep-Now
Record Dates: First submitted 2018-02-09; First posted 2018-02-23 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Cancer of Prostate; Insomnia
MeSH Terms: conditions — Prostatic Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week aerobic exercise and cognitive-behavioral therapy (Experimental): 12-week aerobic exercise, two times per week, and cognitive-behavioral therapy for insomnia in total four sessions
  Interventions: Behavioral: 12-week aerobic exercise and cognitive-behavioral therapy
- Control group (No Intervention): Patients assigned to the control group will receive usual care

INTERVENTIONS:
Behavioral: 12-week aerobic exercise and cognitive-behavioral therapy — 12-week intervention of aerobic exercise training and four session of cognitive-behavioral therapy
  Arms: 12-week aerobic exercise and cognitive-behavioral therapy

SUMMARY:
This study of a randomized controlled trial aims to evaluate the feasibility of a 12-week sleep program and the randomized controlled trial research procedure. In total 20 participants will be recruited and randomized to the intervention or control group.

DETAILED DESCRIPTION:
This feasibility study of a randomized controlled trial, aims to evaluate the feasibility of a 12-week sleep program consisting on aerobic exercise and cognitive-behavioral therapy. In this study the investigators wish to evaluate the program as well as the randomized controlled trial research procedure.

In total 20 participants will be recruited and randomized to either the intervention group (n=10) or control group (n=10).The intervention group will participate in two exercise sessions each week and four sessions based on cognitive-behavioral therapy for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Receiving treatment with androgen deprivation therapy or in combination with chemotherapy
* Insomnia
* Over 18-yers old
* Understand oral and written Danish
* Written informed consent

Exclusion Criteria:

* Medical assessment that does not allow aerobic exercise
* Severe cognitive problems
* Night work during the interventions period
* Exercise training more than three times a week

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Sleep | Change from baseline sleep at 12 weeks
  Measured by actigraphy, to investigate change in sleep from baseline to 12 weeks and the difference in change between intervention - and the control group

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline, 12-weeks
  Measured by watt max test, to investigate change from baseline to 12 weeks and the difference in change between intervention and the control group
Fatigue | Baseline, 12 weeks, 6 month
  Measured by the multidimensional fatigue inventory, to investigate change in fatigue from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Physical activity | Baseline, 12 weeks, 6 month
  Measured by the Physical activity Questionnaire to investigate change in physical activity from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Depression | Baseline, 12 weeks, 6 month
  Measured by the Patient Health Questionnaireto, to investigate change in depression from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Anxiety | Baseline, 12 weeks, 6 month
  Measured by the Generalized Anxiety Disorder Questionnaireto, to investigate change in anxiety from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Stress | Baseline, 12 weeks, 6 month
  Measured by Perceived Stress Scale to investigate change in stress from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Quality of life | Baseline, 12 weeks, 6 month
  Measured by European Organization for Research and Treatment Cancer, to investigate change in quality of life from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Sleep quality | Baseline, 12 weeks, 6 month
  Measured by Pittsburgh Sleep Quality Index, to investigate change in sleep quality from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Sleep pattern | Baseline, 12 weeks, 6 month
  Measured by a sleep diary, to investigate change in sleep pattern from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Insomnia | Baseline, 12 weeks, 6 month
  Measured by Insomnia Severity Index, to investigate change in insomnia from baseline to 12 weeks and 6 months follow up and the difference in change between intervention - and the control group
Physical activity | Baseline, 12 weeks
  Measured by actigraphy, to investigate change in physical activity from baseline to 12 weeks and the difference in change between intervention - and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, PhD, Dr.Med, Principal Investigator — Danish Cancer Society Research Center; Katrine Løppenthin, PhD, Principal Investigator — Danish Cancer Society Research Center
Locations (1):
- Oncology Department, Næstved, Denmark